CLINICAL TRIAL: NCT03054792
Title: Molecular-Functional Imaging of Hypoxia in Childhood Sarcomas: Feasibility Steps Toward Personalized Medicine.
Brief Title: Molecular-Functional Imaging of Hypoxia in Childhood Sarcomas
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andrea Doria, Radiologist, Scientist, Research Director, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000049533
Record Dates: First submitted 2017-01-26; First posted 2017-02-16 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Rhabdomyosarcoma; Non-Rhabdo. Soft Tissue Sarcoma
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BOLD- DW- MRS (Experimental): Blood Oxygen Level Dependent [BOLD], Diffusion-Weighted [DW] MRI, MR Spectroscopy [MRS]
  Interventions: Diagnostic Test: Blood Oxygen Level Dependent [BOLD] MRI; Diagnostic Test: Diffusion-Weighted [DW] MRI; Diagnostic Test: Magnetic Resonance Spectroscopy [MRS]

INTERVENTIONS:
Diagnostic Test: Blood Oxygen Level Dependent [BOLD] MRI — BOLD is a non-invasive T2*-weighted MRI technique that is sensitive to the microvascular deoxyhemoglobin concentration. BOLD has the potential to monitor changes in tissue oxygenation in response to a gas breathing challenge to induce contrast.
Diagnostic Test: Diffusion-Weighted [DW] MRI — DW MRI is a non-invasive technique that provides quantitative biophysical information about the movement of water in tissues and reflects the anisotropy of normal and pathologic cells
Diagnostic Test: Magnetic Resonance Spectroscopy [MRS] — MRS is a non-invasive imaging technique that enables the generation of spectral profiles of low molecular weight metabolites that reflect status of a tissue

SUMMARY:
This study will test the feasibility of using novel/existing imaging technologies focused on hypoxia measurements to determine "response to therapy" in pediatric soft tissue sarcomas as a pilot study. Specifically, the investigators will compare the sensitivity of Blood Oxygen Level Dependent [BOLD], Diffusion-Weighted [DW] MRI and Magnetic Resonance Spectroscopy (MRS) with that of conventional MRI to detect measurement changes between the start and completion of neoadjuvant therapy ("response to therapy") in children and adolescents (6-18 years) with suspicion of sarcoma tumors. Clinicians and scientists may use results of the proposed hypoxia-imaging surrogate markers to adjust/modify therapeutic schemes to patients on a personalized basis.

ELIGIBILITY:
Inclusion Criteria:

* Referred with a confirmed or suspected sarcoma tumor (rhabdomyosarcoma [RMS] or non-rhabdomyomatous sarcoma) presenting with an extra-osseous component;
* Candidate for neoadjuvant therapy that will consist of standard systemic chemotherapy with or without radiation therapy

Exclusion Criteria:

* Patients with general contraindications for an MRI scan (metal foreign body, pacemaker, inability to tolerate an examination without sedation);
* Patients with a known immunodeficiency/sickle cell disease/collagen vascular disease/another malignancy;
* Patients with no clinical indication for neoadjuvant therapy prior to surgery;
* Patients with chronic pulmonary disease;
* Patients with other diagnosis confirmed after initial suspicion of RMS or non-RMS.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with response to therapy | 1 year
  Response will be assessed by measurements of tumor volume, percentage of BOLD signal changes, percentage of tumor necrosis, apparent diffusion coefficient, concentration of high-energy and low-energy phosphates in tumor.

SECONDARY OUTCOMES:
Associations between post-neoadjuvant therapy imaging measurements and surgical / histochemical outcomes in the residual tumor. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared with other researchers